CLINICAL TRIAL: NCT06083103
Title: Contribution of PET/MRI in Locally Advanced Cervical Cancer
Brief Title: Contribution of PET/MRI in Locally Advanced Cervical Cancer (ATICC)
Acronym: ATICC
Status: Recruiting | Type: Observational
Sponsor: Centre Paul Strauss (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-013; 2023-A00743-42 (Other: ID-RCB Number)
Record Dates: First submitted 2023-10-06; First posted 2023-10-13 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 18-FDG PET-MRI — For this trial, 18-FDG PET-MRI will be conducted directly after PET-CT using a single dose of radiotracer

SUMMARY:
[18 F]fluorodeoxyglucose (18F-FDG) positron emission tomography-magnetic resonance imaging (PET/MRI) is a new hybrid imaging tool that has recently arrived in oncology, and is particularly promising. Its usefulness seems obvious in certain tumor types, but its place in the staging of cervical cancers has never been explored in a prospective trial to our knowledge.

Previously, a comparative retrospective study from 2009 found a better sensitivity of PET fused to diagnostic MRI images compared to PET/CT (positron emission tomography/computed tomography) in the detection of metastatic lymph nodes (54 and 44% respectively). It was an a posteriori fusion of images, from images acquired by PET-CT.

DETAILED DESCRIPTION:
This monocentric, prospective trial aims at comparing performances of 18F-FDG PET/MRI versus standard PET/CT in the detection of lymph node metastases in cervical cancer patients. Specificity and sensitivity of both exams will be compared at one timepoint, during the PET/CT prescribed in routine care for assessment of extension. PET/MRI will be conducted directly after PET/CT and a unique dose of 18F-FDG radiotracer will be used for both exams.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 years old and over
* Patients with presumed cervical cancer of stages IB2 to IVA based on clinical data and pelvic MRI, undergoing pre-treatment assessment.
* For women of childbearing potential : Adequate contraception throughout study participation.

Note : enrollment in a concomitant clinical trial is authorized

Exclusion Criteria:

* Oncological history that could possibly interfere with imaging results interpretation, apart from cervical cancer
* Extra-nodal metastasis clinically or radiologically proven before study participation
* Contraindication to MRI or injection of contrast agents containing gadolinium
* Contraindication to lumbo-aortic lymphadenectomy
* Persons deprived of liberty
* Minor or patients placed under guardianship or supervision
* Patient under judicial protection
* Patient unable to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with presumed cervical cancer of stages IB2 to IVA based on clinical data and pelvic MRI, undergoing pre-treatment assessment.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Compare performances of PET/MRI and PET/CT in the detection of lumbar aortic lymph node metastases in cervical cancer patients with tumors graded IB2 to IVA stage | Up to 3 months
  Performances in terms of sensitivity

SECONDARY OUTCOMES:
Compare performances of PET/MRI and PET/CT in the detection of lymph node metastases in cervical cancer patients with tumors graded IB2 to IVA stage, outside of lumbar aortic region | Up to 3 months
  Performances in terms of sensitivity
Compare performances PET/MRI and para-aortic lymphadenectomy in the detection of lumbar aortic lymph node metastases in cervical cancer patients | Up to 3 months
  Lumbar/aortic lymph nodes detection with each exams

CONTACTS AND LOCATIONS:
Overall Officials: Éric OUVRARD, MD, Study Chair — Institut de cancérologie Strasbourg Europe
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Picardi M, Cavaliere C, Della Pepa R, Nicolai E, Soricelli A, Giordano C, Pugliese N, Rascato MG, Cappuccio I, Campagna G, Cerchione C, Vigliar E, Troncone G, Mascolo M, Franzese M, Castaldo R, Salvatore M, Pane F. PET/MRI for staging patients with Hodgkin lymphoma: equivalent results with PET/CT in a prospective trial. Ann Hematol. 2021 Jun;100(6):1525-1535. doi: 10.1007/s00277-021-04537-5. Epub 2021 Apr 28. PMID 33909101
- [Background] Lu XR, Qu MM, Zhai YN, Feng W, Gao Y, Lei JQ. Diagnostic role of 18F-FDG PET/MRI in the TNM staging of breast cancer: a systematic review and meta-analysis. Ann Palliat Med. 2021 Apr;10(4):4328-4337. doi: 10.21037/apm-20-2555. Epub 2021 Apr 12. PMID 33894709
- [Background] Crimi F, Spolverato G, Lacognata C, Garieri M, Cecchin D, Urso ED, Zucchetta P, Pucciarelli S, Pomerri F. 18F-FDG PET/MRI for Rectal Cancer TNM Restaging After Preoperative Chemoradiotherapy: Initial Experience. Dis Colon Rectum. 2020 Mar;63(3):310-318. doi: 10.1097/DCR.0000000000001568. PMID 31842163
- [Background] Kim SK, Choi HJ, Park SY, Lee HY, Seo SS, Yoo CW, Jung DC, Kang S, Cho KS. Additional value of MR/PET fusion compared with PET/CT in the detection of lymph node metastases in cervical cancer patients. Eur J Cancer. 2009 Aug;45(12):2103-9. doi: 10.1016/j.ejca.2009.04.006. Epub 2009 May 4. PMID 19403303